CLINICAL TRIAL: NCT06241287
Title: Better Living With Non-memory-led Dementia: a Randomised Controlled Trial of a Web-based Caregiver Educational Programme
Brief Title: BELIDE: Better Living With Non-memory-led Dementia
Acronym: BELIDE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 8545/007
Record Dates: First submitted 2024-01-03; First posted 2024-02-05 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia | interventions — Waiting Lists

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: It is not possible to blind the individual participants in this trial, but the individuals who will be analysing data or overseeing trial including health economists, co- investigators and trial statistician will remain blind until the blinded analysis detailed in the Statistical Analysis Plan has been conducted and reported to the trial team. The exception will be one of the co-investigators leading the process analysis.Unblinding will be performed following procedures outlined in NWORTH SOPs.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group will receive the Better Living with Non-memory led Dementia programme, an 8-week duration 6-module educational programme covering the following topics: 1) Welcome to the programme and what to expect from it; 2) Understanding the disease; 3) How to provide better support for the person with dementia; 4) How to look after the caregiver's own mental health; 5) Where to find additional sources of support, and 6) An introduction to the value of support groups.
  Interventions: Behavioral: Better Living with Non-memory led Dementia programme
- Control group (Other): The waiting list control group will receive signposting to the publicly available Rare Dementia Support website (https://www.raredementiasupport.org/) and any kind of support the participants may already being receiving (e.g. psychological support, online information, support groups, etc). This a wait list study where the control group will be given access to the intervention ́s educational modules and material after the individuals' last point of data collection.
  Interventions: Other: Waiting list

INTERVENTIONS:
Behavioral: Better Living with Non-memory led Dementia programme — an 8-week duration 6-module educational programme covering the following topics: 1) Welcome to the programme and what to expect from it; 2) Understanding the disease; 3) How to provide better support for the person with dementia; 4) How to look after the caregiver's own mental health; 5) Where to find additional sources of support, and 6) An introduction to the value of support groups. At the end of modules 2, 3, and 4, participants will be asked to complete a real-life task to put in practice skills learned in the specific module (e.g., approaching a friend and explaining the disease in lay terms). The first session (onboarding) will be facilitated via Zoom by one of the members of the research team. Up to 3 total interactions between facilitators and participants will be offered to support participants' engagement with the programme. All course modules will be printable using the pdf download button on the programme's page.
  Arms: Intervention group
Other: Waiting list — Signposting individuals to the publicly available Rare Dementia Support website. The control group will further receive access to the Better Living with Non-memory led Dementia programme after completing the collection of measures at 6 months.
  Arms: Control group

SUMMARY:
Around 48 million people worldwide 1 live with dementia, of whom 3.9 million start with symptoms before the age of 65 (young-onset dementia). Most of the people presenting with young-onset dementia and some people with later onset dementia develop non-memory led dementias such as the atypical forms of Alzheimer ́s disease (AD)or frontotemporal dementia (FTD). Despite the proven benefits of educational programmes and skill training for caregivers, families of people with non-memory led dementias encounter fewer opportunities to receive this type of support. This is a significant gap in care considering that many people with young-onset non-memory led dementia are in their 50s or early 60s, which carries additional challenges about employment, financial stability, and childcare responsibilities. Finding suitable information and resources is less likely due to the lower prevalence of these phenotypes, their consequent geographical spread, and their atypical symptoms. Caregivers demands for more phenotype-specific support suggest that tailored provision of education and training is a gap in the provision of care in these types of dementia.

The aim of this study is to:

1. Determine the effectiveness of the Better Living with Non-memory Dementia educational programme for caregivers in improving psychological outcomes [WS1]; and
2. Conduct a mixed methods process analysis to elucidate mechanisms of change, barriers and facilitators to access and implementation as well as perceived benefits and costs [WS2].

The design is a randomised waiting list control trial with an 8-week intervention and 6-month follow-up comparing intervention to standard care with embedded process analysis. The intervention comprises a virtual onboarding session with a facilitator, 6 learning modules (including module-end real-life tasks to put skills into practice) and up to two further virtual check-in sessions with the facilitator. Intervention adaptation, adaptation to design and selection of primary outcome measures was based on feasibility work.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (18+) who self-identify as an unpaid carer (partners, children, friends, etc.) of someone with PPA, PCA or bvFTD who is not living in a full-time care facility.
2. The care recipient must have a confirmed diagnosis of dementia (through self-report of the carer, to reflect the 'real world' application of the intervention).
3. Able to give informed consent.
4. Good comprehension of written English.
5. Access to the internet.

Exclusion Criteria:

1. Carers of people living with dementia in full-time care facility.
2. Carers of people with severe dementia in terms of large impact on activities of daily living.
3. Carers of individuals with any form of dementia other than PPA, PCA, or bvFTD. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 238 (Estimated)
Dates: Start 2024-01-29 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire (PHQ 9) | 8 weeks
  Are Patient Health Questionnaire (PHQ 9) scores significantly decreased in caregiver participants allocated to receive the intervention compared to participants allocated to a waiting list control group.
  Scores can range from 0 to 27. Higher score mean worse outcome.

SECONDARY OUTCOMES:
Perceived Stress Scale (PSS) | 8 weeks
  Measures perceived stress.
  Scores can range from 0 to 40. Higher score mean worse outcome.
Caregiver Self-efficacy Scale (CSES-8). Scores can range from 1 to 10. Higher score mean better outcome. | 8 weeks
  Measures perceived caregiver self-efficacy
ICEpop Capability measure for adults (ICECAP-A) | 8 weeks
  Measures capability for the general adult population for use un economic evaluation.
  Scores can range from 5 to 25. Higher score mean better outcome.
Quality of Carer-Patient relationship (QCPR) | 8 weeks
  Measures the quality of the carer patient relationship.
  Scores can range from 14 to 70. Higher score mean better outcome.
Health related quality of life (EQ5D5L) | 8 weeks
  EuroQol Group tool to measure quality of life related to health outcomes.
  Scores can range from 5 to 25. Higher score mean better outcome.

OTHER OUTCOMES:
Qualitative interviews | week 8 and 24
  Semi-structured interviews will be conducted with a subset of participants who complete the BELIDE intervention, to explore their experiences of using the online tool, perceived benefits or challenges, and its impact on their caregiving role.

CONTACTS AND LOCATIONS:
Locations (1):
- University College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Suarez-Gonzalez A, Brotherhood E, John A, Hayes O, Rossi-Harries S, Zimmermann N, Mansfield V, Brand A, Hoare Z, Fitzsimmons D, Cullen K, Crutch S, Stott J. Better Living with Non-memory-led Dementia: study protocol for a randomised controlled trial of a web-based caregiver educational programme (BELIDE trial). BMJ Open. 2025 Sep 5;15(9):e102518. doi: 10.1136/bmjopen-2025-102518. PMID 40912705